CLINICAL TRIAL: NCT02948218
Title: Multi-center Clinical Research of Acupuncture Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCRATKO
Record Dates: First submitted 2016-10-16; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Shanghai Longhua hospital (Active Comparator): Acupuncture treatments will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.
  Interventions: Device: Acupuncture treatment
- Shanghai Guanghua hospital (Active Comparator): Acupuncture treatments will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.
  Interventions: Device: Acupuncture treatment
- Huadong hospital of Fudan University (Active Comparator): Acupuncture treatments will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.
  Interventions: Device: Acupuncture treatment
- Shanghai Yueyang Integrated hospital (Active Comparator): Acupuncture treatments will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.
  Interventions: Device: Acupuncture treatment

INTERVENTIONS:
Device: Acupuncture treatment — Acupuncture treatment will be the Traditional Chinese Medicine type. Acupuncture 3 times per week, 4 weeks is one treatment period. Every patient will be given 3 treatment period.

SUMMARY:
Knee osteoarthritis (KOA) is a major public health problem among the elderly and is associated with considerable disability. A recent analysis of data indicated that about 35% of women and men aged 60 years and above had radiographic knee OA.Despite the high prevalence rate of OA, the treatment of OA is far from satisfactory. Acupuncture may be a promising treatment option for knee OA due to the effectiveness of the pain relief and the rarity of adverse effects. In order to get some more reliable data to confirm acupuncture effectiveness on KOA, a long-term follow up interventional study will be started to confirm the effects of long term for acupuncture treatment.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a major public health problem among the elderly and is associated with considerable disability. A recent analysis of data from the National Health and Nutrition Examination Survey III indicated that about 35% of women and men aged 60 years and above had radiographic knee OA. Although the cause of OA can be many factors, such as previous injury, abnormal limb development and so on, its main symptom is a complex chronic pain condition. Previous studies have demonstrated central sensitization in OA patients. Despite the high prevalence rate of OA, the treatment of OA is far from satisfactory. Acupuncture could be a promising treatment option for knee OA due to the effectiveness of the pain relief and the rarity of adverse effects. In order to get some more reliable data to confirm acupuncture effectiveness on KOA, a long-term follow up interventional study with clear design, standard criteria, control group, will be started to confirm the effects of long term for acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients who have knee OA diagnosed according to the American College of Rheumatology classification criteria (with at least one osteophyte in the tibiofemoral joint and with a Kellgren-Lawrence grade of more than 2).
* Male and female patients who have had a history of moderate or greater knee pain of more than 3 months' duration and have reported moderate or greater, clinically significant, knee pain during most days of the last month before the interview.
* Male and female patients who have given their consent to participate in the study.
* Patients will be selected among those who are not on the waiting list for total knee arthroplasty by the traumatology unit of our hospital.

Exclusion Criteria:

* Patients with any of the following will be excluded from the study: a history of any secondary OA associated with any systemic arthropathy (i.e., rheumatoid arthritis or gouty arthritis);
* Any knee treatment with steroids, methotrexate, or azathioprine; recent traumatisms caused by acupunctured insertion;
* A history of bleeding disorders or any disease related to acupuncture contraindications;
* A history of any knee injection in the previous 6 months (e.g., cortisone and hyaluronic acid); a history of morphine or morphine derivative use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 12 weeks
  Visual analogue scale assessed for 12 weeks

SECONDARY OUTCOMES:
Western Ontario and McMaster university of orthopedic index | 12weeks
  Western Ontario and McMaster university of orthopedic index assessed for 12 weeks.
Lequesne index | 12 weeks
  Lequesne index assessed for 12 weeks.
Adverse Event | 12 weeks
  Adverse Event assessed for 12 weeks.
The Medical Outcomes Study short form health survey-36 | 12 weeks
  The Medical Outcomes Study short form health survey-36 assessed for 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Ph.D, M.D, Study Director — Shanghai Longhua Hospital
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data (IPD) available

REFERENCES:
- [Result] Ho-Pham LT, Lai TQ, Mai LD, Doan MC, Pham HN, Nguyen TV. Prevalence of radiographic osteoarthritis of the knee and its relationship to self-reported pain. PLoS One. 2014 Apr 10;9(4):e94563. doi: 10.1371/journal.pone.0094563. eCollection 2014. PMID 24722559
- [Result] Nguyen US, Zhang Y, Zhu Y, Niu J, Zhang B, Felson DT. Increasing prevalence of knee pain and symptomatic knee osteoarthritis: survey and cohort data. Ann Intern Med. 2011 Dec 6;155(11):725-32. doi: 10.7326/0003-4819-155-11-201112060-00004. PMID 22147711
- [Result] Hochman JR, Davis AM, Elkayam J, Gagliese L, Hawker GA. Neuropathic pain symptoms on the modified painDETECT correlate with signs of central sensitization in knee osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1236-42. doi: 10.1016/j.joca.2013.06.023. PMID 23973136
- [Result] Finan PH, Buenaver LF, Bounds SC, Hussain S, Park RJ, Haque UJ, Campbell CM, Haythornthwaite JA, Edwards RR, Smith MT. Discordance between pain and radiographic severity in knee osteoarthritis: findings from quantitative sensory testing of central sensitization. Arthritis Rheum. 2013 Feb;65(2):363-72. doi: 10.1002/art.34646. PMID 22961435
- [Result] Berman BM, Lao L, Langenberg P, Lee WL, Gilpin AM, Hochberg MC. Effectiveness of acupuncture as adjunctive therapy in osteoarthritis of the knee: a randomized, controlled trial. Ann Intern Med. 2004 Dec 21;141(12):901-10. doi: 10.7326/0003-4819-141-12-200412210-00006. PMID 15611487
- [Result] Hinman RS, McCrory P, Pirotta M, Relf I, Forbes A, Crossley KM, Williamson E, Kyriakides M, Novy K, Metcalf BR, Harris A, Reddy P, Conaghan PG, Bennell KL. Acupuncture for chronic knee pain: a randomized clinical trial. JAMA. 2014 Oct 1;312(13):1313-22. doi: 10.1001/jama.2014.12660. PMID 25268438
- [Result] White A, Hayhoe S, Hart A, Ernst E. Adverse events following acupuncture: prospective survey of 32 000 consultations with doctors and physiotherapists. BMJ. 2001 Sep 1;323(7311):485-6. doi: 10.1136/bmj.323.7311.485. No abstract available. PMID 11532840